CLINICAL TRIAL: NCT06147531
Title: A Clinical Comparison of Cold-stored and Room Temperature-stored Allogeneic Platelet Transfusions in Bleeding Adult Cardiac Surgery Patients - A Randomized Multicentre Pilot Study (PLTS-1 Study)
Brief Title: Delayed Cold-Stored Platelets -PLTS-1
Acronym: PLTS-1
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: University Health Network, Toronto (Other)
Collaborators: Kingston Health Sciences Centre (Other); Canadian Blood Services (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 22-5855
Record Dates: First submitted 2023-10-31; First posted 2023-11-27 (Actual); Last update posted 2025-12-29 (Actual); Status verified 2025-12

CONDITIONS: Platelets; Bleeding; Cardiopulmonary Bypass; Cardiac Surgery
Keywords: Blood Platelets; Cardiac surgical procedure; Blood Preservation/Methods; Blood Preservation/Adverse Effects
MeSH Terms: conditions — Hemorrhage

STUDY DESIGN:
Intervention Model Description: PLTS-1 is a multicentre, randomized, controlled, pilot trial, using a conventional, parallel group, two-armed design at 2 cardiac surgery centres in Canada.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: This will be a blinded randomized trial, with clinical personnel, patients, family members, and outcome assessors blinded to group allocation. Given that the platelets will be different temperatures (but identical in appearance), an unblinded blood bank technologist, who will not have access to the collected study data, will blind the platelets by placing them in an insulated tamper-proof container accompanied by a pair of disposable insulated gloves. The clinician(s) directly handling the product at the time of transfusion will wear the insulated gloves to prevent unblinding (simulations have shown this to be an effective strategy). The platelets will also have blinded study labels and come prepared in identical collection bags.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention Group (Experimental): Patients randomized to the Delayed Cold-Stored Platelet Group will receive ABO-identical buffy-coat platelets (pathogen reduced products) maintained at 22°C for up to 4 days then placed at 4°C for a minimum of 1 day (24 hours), with expiration at 14 days after collection.
  Interventions: Biological: Delayed Cold-Stored Buffy Coat Platelets
- Control Group (Active Comparator): Those randomized to the Room Temperature Platelet Group will receive ABO-identical buffy-coat platelets (pathogen reduced products) maintained at 22°C for up to 7 days (as per current standard of care).
  Interventions: Biological: Room Temperature Buffy Coat Platelets

INTERVENTIONS:
Biological: Delayed Cold-Stored Buffy Coat Platelets — To prepare cold-stored platelets, blood banks will transition conventional room temperature platelets up to 4 days after collection (with agitation) to cold-storage (at 1-6 C without agitation) for a minimum of 1 day (24 hours) and a maximum of 10 days after collection (for a total shelf life of ≤ 14 days after collection). Thus, cold-stored platelets will be produced and stored the same way as room temperature platelets up until their transition to cold-storage, ensuring similar products differing only in storage conditions and expiration date (as cold-stored platelets will have an expiration date beyond the current 5 days for pathogen inactivated platelets or 7 days for bacterially cultured platelets). Pathogen reduced platelets will be used for the pilot study (Canada is transitioning in 2022-23 to pathogen-reduced platelets and one site has already transitioned).
  Arms: Intervention Group
Biological: Room Temperature Buffy Coat Platelets — Room temperature stored platelets are prepared from donor whole blood, which is centrifuged to collect the buffy coat layer containing platelets. Seven ABO matched buffy coats from male and/or female donors are pooled in 280 ml of platelet additive solution and split into a single dose after pathogen inactivation, resulting in a product with a final platelet count of approximately 1300 x 109. Pathogen inactivated platelets (shelf-life of 5 days, with recent Health Canada approval for an extension of the shelf-life to 7 days), will be used as Canada is transitioning in 2022-23 to pathogen-inactivated platelets and one site has already transitioned.
  Arms: Control Group

SUMMARY:
PLTS-1 is a multicentre, randomized, controlled, pilot trial, using a conventional, parallel group, two-armed design at 2 cardiac surgery centres in Canada. The study is designed to assess the feasibility of a future, definitive RCT to determine the non-inferiority of cold-stored platelets compared to conventional platelets with respect to hemostatic effectiveness (total number of allogeneic blood products transfused within 24 hours after CPB), as well as safety.

ELIGIBILITY:
Inclusion Criteria:

Adult (≥18 years old) patients undergoing elective cardiac surgery with CPB will be eligible for inclusion if they are planned to undergo at least moderately complex surgery or have a preoperative platelet count ≤150,000 x106/L (this is a group at high risk of requiring platelet transfusions post-CPB).

Moderately complex index surgery is defined as:

1. repair/replacement of more than one valve;
2. aorta (root/ascending/arch) replacement;
3. any combination of coronary artery bypass grafting, valve repair/replacement, or aorta (root/ascending/arch) replacement; or
4. re-do procedures consisting of a repair or revision of a prior cardiac intervention.

Exclusion Criteria:

Patients will be excluded if cold-stored platelets are not going to be available at the time of surgery or if the patient:

1. has a congenital or acquired hemostatic disorder (including platelet refractoriness due to anti-platelet and anti-human leukocyte antigen [HLA] antibodies) and/or requires specially matched platelets (including patients with anaphylaxis to blood due to Immunoglobulin A [IgA] deficiency),
2. has known contraindications to heparin, thereby excluding cases where non-reversible anticoagulants (i.e. argatroban) are used,
3. is on warfarin or direct oral anticoagulants (dabigatran, rivaroxaban, apixaban or edoxaban) within 3 days prior to surgery,
4. is on antiplatelet drugs within 5 days prior to surgery (excluding acetylsalicylic acid [ASA]),
5. refuses allogeneic blood products,
6. has a known pregnancy,
7. has already enrolled in this study,
8. is enrolled in another interventional clinical trial where routine care and management are altered,
9. has hemodynamic instability defined as critical care admission, vasopressor, or inotrope dependence prior to index surgery, or
10. has pre-operative requirement for, or expected post-operative dependence upon mechanical circulatory support (i.e., intra-aortic balloon pump, ventricular assist device).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Estimated)
Dates: Start 2024-06-05 (Actual); Primary Completion 2026-06 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Feasibility Outcome 1: Adequate Patient Recruitment | through study completion, an average of 1 year.
  Adequate recruitment (defined as ≥ 15% of eligible patients enrolled per centre per month to target consistent levels of enrollment).
Feasibility Outcome 2: Adequate cold-stored platelet supply | through study completion, an average of 1 year.
  Adequate cold-stored platelet supply (defined as appropriate product available at the time of surgery for ≥90% of patients randomized to the cold-stored platelet group).
Feasibility Outcome 3: Adequate clinician adherence to randomization assignment. | through study completion, an average of 1 year.
  Adequate clinician adherence to randomization assignment (defined as >90% of all randomized patients are administered the assigned product).

CONTACTS AND LOCATIONS:
Overall Officials: Justyna Bartoszko, MD, Principal Investigator — University Health Network, Toronto; Jeannie Callum, MD, Principal Investigator — Kingston Health Sciences Centre
Locations (2):
- Canada (2):
  - Kingston Health Sciences Centre, Kingston, Ontario
  - Toronto General Hospital - University Health Network, Toronto, Ontario

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Bartoszko J, Peer M, Grewal D, Ansari S, Callum J, Karkouti K. Delayed cold-stored vs. room temperature stored platelet transfusions in bleeding adult cardiac surgery patients-a randomized multicentre pilot study (PLTS-1). Pilot Feasibility Stud. 2024 Jun 15;10(1):90. doi: 10.1186/s40814-024-01518-z. PMID 38879518